CLINICAL TRIAL: NCT02452450
Title: Ibuprofen and Paracetamol Pharmacokinetic Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Reckitt Benckiser Healthcare (UK) Limited (Industry)
Collaborators: Simbec Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: NL1307
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Healthy Volunteer Study
MeSH Terms: interventions — Ibuprofen; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Ibuprofen lysine (Experimental)
  Interventions: Drug: Ibuprofen Lysine
- Ibuprofen sodium (Experimental)
  Interventions: Drug: Ibuprofen Sodium
- Ibuprofen liquid capsules (Experimental)
  Interventions: Drug: Ibuprofen Liquid Capsules
- Ibuprofen acid (Active Comparator)
  Interventions: Drug: Ibuprofen Acid
- Paracetamol (Active Comparator)
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Ibuprofen Acid
  Arms: Ibuprofen acid
Drug: Ibuprofen Lysine
  Arms: Ibuprofen lysine
Drug: Ibuprofen Sodium
  Arms: Ibuprofen sodium
Drug: Ibuprofen Liquid Capsules
  Arms: Ibuprofen liquid capsules
Drug: Paracetamol
  Arms: Paracetamol

SUMMARY:
The purpose of this study was to determine rates of absorption of Ibuprofen and Paracetamol formulations.

ELIGIBILITY:
Inclusion Criteria:

1. Age: > 18 to < 50 years.
2. Sex: Male and female subjects are eligible for entry.
3. Female subject of child bearing potential with a negative pregnancy test at the screening visit and willing to use an effective method of contraception, if applicable
4. Female subject of non-child bearing potential with negative pregnancy test at the screening visit.
5. Male subject willing to use an effective method of contraception.
6. Status: Healthy volunteers with a body mass index of >18 and <30 kg/m2.
7. Absence of relevant abnormalities in the clinical examination, ECG, drug and safety analysis.
8. Subjects who have given written informed consent

Exclusion Criteria:

1. Pregnant or lactating female subjects.
2. A history of significant disease of any body-system.
3. Any condition that may currently interfere with the absorption, distribution, metabolism or excretion of drugs.
4. A history of allergy or intolerance (including angio-oedema, urticaria, bronchospasm and rhinitis) related to treatment with ibuprofen, aspirin or other non-steroidal anti-inflammatory drugs (NSAIDs), paracetamol, or the excipients of the formulations.
5. A history of peptic or duodenal ulcers or gastro-intestinal bleed or upper gastro-intestinal bleed, or other significant gastro-intestinal disorders.
6. A history of frequent dyspepsia, e.g., heartburn or indigestion.
7. A history of migraine.
8. A history of psychotic illness, attempted suicide or parasuicide.
9. Current smokers and ex-smokers who have smoked within 6 months.
10. A history of drug abuse (including alcohol).
11. High consumption of stimulating drinks
12. Those with positive drugs of abuse screen including alcohol on any occasion throughout the study.
13. Ingestion of a prescribed drug at any time in the 14 days before dosing with study medication (excluding hormonal contraceptives and hormone replacement therapy), or consumption of enzyme inhibitors or inducers during the previous month (such as barbiturates, carbamazepine, erythromycin, phenytoin, etc).
14. Ingestion of an over-the-counter preparation within 7 days before dosing with study medication, including herbal medications, vitamin/fish oil supplements, ibuprofen and other NSAIDs and paracetamol.
15. Donation of blood in quantity in the previous 12 weeks before enrolment into the study
16. Known human immune deficiency virus (HIV) positive status, or a positive viral serology screen.
17. Topical use of ibuprofen within 7 days before dosing with study medication
18. Those previously randomised into this study.
19. Employee at study site.
20. Partner or first degree relative of the investigator.
21. Those with an ibuprofen level > 10 ng/ml as determined at pre-study screening visit 2 (Part 2 (Pivotal Phase) of the study only).
22. Those who are unwilling to consume gelatin of animal origin (Part 2 (Pivotal Phase) of the study only).
23. Those who have participated in a clinical trial in the previous 12 weeks
24. Those unable in the opinion of the Investigator to comply fully with the study requirements.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2014-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Time to the maximum concentration (Cmax) of the reference Ibuprofen | 0-4hr
Time to the first extrapolated non-zero concentration (Tlag) | 0-4hr
Time to the maximum concentration (Tmax) | 0-4hr

SECONDARY OUTCOMES:
Time to the lower therapeutic level reaching at least 5 µg/ml (T5.0) for ibuprofen and paracetamol | 0-4hr
Time to the mid therapeutic level reaching at least 8.4 µg/ml (T8.4) for ibuprofen and 10 µg/ml (T10.0) for paracetamol | 0-4hr
Time to the higher therapeutic level reaching at least 10.0 µg/ml (T10.0) for ibuprofen and 20 µg/ml (T20.0) for paracetamol | 0-4hr
Partial area under the curve (AUCs) at each nominal blood sampling time-point | 0-4hr
The area under the curve up to the median Tmax for the ibuprofen reference product (AUCTmaxRef) | 0-4hr
The plasma concentration at each planned nominal time-point (Cn) | 0-4hr
The maximum plasma concentration (Cmax) | 0-4hr

REFERENCES:
- [Derived] Miles L, Hall J, Jenner B, Addis R, Hutchings S. Predicting rapid analgesic onset of ibuprofen salts compared with ibuprofen acid: Tlag, Tlow, Tmed, and a novel parameter, TCmaxRef. Curr Med Res Opin. 2018 Aug;34(8):1483-1490. doi: 10.1080/03007995.2018.1466697. Epub 2018 Apr 27. PMID 29667449